CLINICAL TRIAL: NCT04892771
Title: Post-healing Follow-up Study in People With Remission of a Diabetic Foot Ulcer
Acronym: Pied-REM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0027
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Diabetic Foot
Keywords: Diabetic foot ulcer; Recurrence; Prevention; Remission; Follow-up; Multidisciplinary team
MeSH Terms: conditions — Diabetic Foot; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Patients who have honored two consultations per year for two years.
- Control group: Patients who have not honored two consultations per year for two years.

SUMMARY:
To evaluate the benefit of multidisciplinary specific follow-up of patients with a healed diabetic foot ulcer at the rate of two annual consultation on wound recurrence.

DETAILED DESCRIPTION:
Diabetic foot ulcer is a major world health problem with a very high recurrence rate, 50% at two years.

The main causes of diabetic foot ulcer recurrence are inadequate footwear, lack of podology care and lack of self-care. International recommendations call for regular podological monitoring to prevent recurrence of diabetic foot ulcer.

The "remission foot" consultation assesses recommended items and is offered to any healed patient at the rate of two annual visit.

A retrospective study on multidisciplinary specific follow-up may show a real efficacity on recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 1 ou type 2 diabetes followed-up in Centre Hospitalier Sud Francilien,
* Discharge from hospital for diabetic foot ulcer between 2017 and 2019 and post-healing follow-up for two years,
* 18 years of âge or older,
* Person not deprived of liberty,
* person who was informed of and did not object to the study.

Exclusion Criteria:

- Person refusing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diabetic foot ulcer healed who were followed-up in CHSF. All these patients have a high podological risk.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Number of wound | At 2 years
  Diabetic foot ulcer recurrence

SECONDARY OUTCOMES:
Hospitalisation | At 2 years
  Days of hospitalisation for diabetic foot ulcer
Number of visits to the pedicure | At 2 years
  Podology follow-up
Adequate footwear | At 2 years
  Wearing of adequate shoes

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Netten JJ, Price PE, Lavery LA, Monteiro-Soares M, Rasmussen A, Jubiz Y, Bus SA; International Working Group on the Diabetic Foot. Prevention of foot ulcers in the at-risk patient with diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:84-98. doi: 10.1002/dmrr.2701. PMID 26340966
- [Background] Bus SA, van Netten JJ, Lavery LA, Monteiro-Soares M, Rasmussen A, Jubiz Y, Price PE; International Working Group on the Diabetic Foot. IWGDF guidance on the prevention of foot ulcers in at-risk patients with diabetes. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:16-24. doi: 10.1002/dmrr.2696. No abstract available. PMID 26334001
- [Background] Bus SA, Waaijman R, Arts M, de Haart M, Busch-Westbroek T, van Baal J, Nollet F. Effect of custom-made footwear on foot ulcer recurrence in diabetes: a multicenter randomized controlled trial. Diabetes Care. 2013 Dec;36(12):4109-16. doi: 10.2337/dc13-0996. Epub 2013 Oct 15. PMID 24130357
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678